CLINICAL TRIAL: NCT03771235
Title: Online Mindfulness-based Tic Reduction: Development and Testing (Phase Two)
Brief Title: Online Mindfulness-based Tic Reduction (Phase Two)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bowdoin College (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hannah Reese, Assistant Professor, Bowdoin College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-30
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Tourette Syndrome; Persistent Tic Disorder
Keywords: Tourette Syndrome; Tic Disorder; Online; Adults; Mindfulness; Therapy
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Coping Skills

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Intervention for Tics (Experimental): 8-week group-based mindfulness-based program
  Interventions: Behavioral: Mindfulness-based Intervention for Tics
- Tic Information and Coping Strategies (Active Comparator): 8-week group-based educational and supportive therapy program
  Interventions: Behavioral: Tic Information and Coping Strategies

INTERVENTIONS:
Behavioral: Mindfulness-based Intervention for Tics — Psychological intervention that focuses on cultivating awareness of urges to tic and developing a different relationship to those urges through meditation and other mindfulness practices.
  Arms: Mindfulness-based Intervention for Tics
Behavioral: Tic Information and Coping Strategies — Psychological Intervention that focuses on learning more about tics, practicing a range of strategies for coping with tics (e.g., relaxation, effective communication), and discussing challenges commonly experienced by individuals with tics.
  Arms: Tic Information and Coping Strategies

SUMMARY:
Tourette Syndrome (TS) and Persistent Tic Disorder (PTD) are chronic and potentially disabling neurobiological conditions. Although a range of pharmacological and psychosocial treatments exists, a significant number of individuals either do not respond to the current treatments or find them unacceptable. Thus, it is essential that researchers continue to develop and test novel treatment approaches.

In this randomized controlled trial the investigators will compare two different online group-based interventions for tics: a mindfulness-based program (Mindfulness-based Intervention for Tics (MBIT), and a psychoeducational and supportive therapy program (Tic Information and Coping Strategies (TICS)). The purpose of this study is to determine which intervention is more helpful for adults with a tic disorder.

ELIGIBILITY:
Inclusion Criteria:

1. be 18 years of age or older,
2. possess a primary diagnosis of Tourette Syndrome or Persistent Tic Disorder,
3. be fluent in English
4. reside in the United States,
5. either not be taking any tic suppressant medication or other psychotropic medication or be at a stable dose for 8 weeks prior to the baseline assessment and throughout the study

Exclusion Criteria:

1. be receiving concurrent psychotherapy for the duration of the study
2. have prior extensive experience with mindfulness and/or meditation and
3. have another medical or psychological condition that would prevent the individual from fully engaging in the study or require a higher level of care (e.g., suicidality).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Change in Yale Global Tic Severity Scale (YGTSS) Total Tic Severity Score | Screening, Week 0, Week 9, Week 13, Week 35
  Clinician-rated measure of tic severity

SECONDARY OUTCOMES:
Clinical Global Impressions Scale | Weeks 0, 9, 13, 35
Adult Tic Questionnaire | Weeks 0, 9, 13, 35
Yale-Brown Obsessive Compulsive Scale | Weeks 0, 9, 13, 35
Attention-Deficit Hyperactivity Rating Scale | Weeks 0, 9, 13, 35
Depression Anxiety Stress Scale | Weeks 0, 9, 13, 35
Premonitory Urge to Tic Scale | Weeks 0, 9, 13, 35
Tic Rating Form | Weeks 1-8
Problem Rating Form | Weeks 1-8
Patient Health Questionnaire-9 | Weeks 0, 9, 13, 35
Work and Social Adjustment Survey | Weeks 0, 9, 13, 35
Five Facet Mindfulness Questionnaire | Weeks 0, 4, 8, 9, 13, 35
Credibility and Expectancy Questionnaire | Week 3
Patient Satisfaction Questionnaire | Week 9
Self Compassion Scale | Weeks 0, 9, 13, 35
Affective Reactivity Index | Weeks 0, 9, 13, 35
Brief Irritability Test | Weeks 0, 9, 13, 35

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Reese, Ph.D., Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - Bowdoin College, Brunswick, Maine
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT03771235/Prot_000.pdf